CLINICAL TRIAL: NCT04168281
Title: Watchful Observation of Patients With Limited Small Cell Lung Cancer Instead of the PCI - Prospective, Multi-center One-arm Study
Brief Title: Watchful Observation of Patients With LD-SCLC Instead of the PCI
Acronym: PCILESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sergiusz Nawrocki (Other)
Responsible Party: Sponsor-Investigator, Sergiusz Nawrocki, Head of Oncology Dept., University of Warmia and Mazury in Olsztyn
Organization: University of Warmia and Mazury in Olsztyn (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LD-SCLC_PCI
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: deescalation of treatment - watchful observation instead of Whole Brain Irradiation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PCI- free after response to radical chemoradiotherapy (Experimental): Patients with no metastases will be followed-up with MRI: at the qualifying visit before MRI-1, and then every 6 months +/- 2 weeks), the patients will have a cognitive examination performed using dedicated neuropsychological tests and QoL assessment using the QLQ-C30 questionnaire. The tests will be conducted in the following order: California verbal learning test (CVLT) with a delay of 15 min, Color connection test (CTT), CVLT (after delay), Benton visual memory test (BNRT), Verbal fluency test by the certified psychologist.
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — instead of PCI patients will be followed-up with MRI

SUMMARY:
Prophylactic cranial irradiation (PCI) is a current standard of care after confirmed response to radical chemoradiotherapy for limited disease small cell lung cancer (LD-SCLC). This standard is mostly based on results of old randomized studies when brain imaging with magnetic resonance (MRI) was not available. Survival benefit of PCI in extended SCLC was recently challenged by results of randomized phase III study from Japan. We propose to carefully follow LD-SCLC patients with MRI instead of PCI in order to apply modern brain irradiation [stereotactic radiotherapy (SRT) in eligible patients or whole brain radiation therapy (WBRT)] to patients who develop metastases and to eliminate long terms neurocognitive deficits caused by PCI in patients who would never develop brain metastases.

Methods and analysis This is a prospective multi-centre one-arm trial. A total of 80 patients diagnosed with LD-SCLC after confirmed response to standard of care radical chemoradiotherapy will be enrolled. Patients will be followed-up by brain MRI every 3 months up to 3 years. Neurocognitive function tests will be performed at baseline and after 12 and 24 months. Patients who develop brain metastases during observation will be irradiated. In case of limited number and volume of metastases SRT will be offered to patients; others will be treated with WBRT. The primary endpoint of the trial is overall survival. We have assumed that our approach will not compromise overall survival of treated patients. 2-year survival will be at least 50% in our trial compared to 36% for a group of 138 patients LD-SCLC from our institution treated in 2003-2006 with radical chemoradiotherapy and PCI. The secondary endpoints were designed to asses the risk of developing brain metastases without PCI; to assess the efficacy of radiotherapy of early detected brain metastases, including the feasibility and efficacy of SRT; to assess neurocognitive functions and QoL in the studied cohort. QLQ-C30 questionnaire and the California Verbal Learning Test (CVLT), Color connection test (CTT), Benton visual memory test (BNRT) and Verbal fluency test (VFT) will be carried out by the certified psychologist.

Ethics and dissemination The trial received ethical approval from the local medical university Bioethical Review Board (Komisja Bioetyczna Collegium Medicum Uniwersytet Warmińsko-Mazurski w Olsztynie). The results of the trial will be disseminated through peer-reviewed publications and conference presentations.

DETAILED DESCRIPTION:
Patients with diagnosed LD-SCLC, after radical treatment with remission or at least a good response after radical therapy, will be eligible for the study. Patients would have had radical radiotherapy to the chest with chemotherapy according to current international guidelines and institutional protocols. A detailed medical history will be collected regarding SCLC and comorbidities. During the qualification visit, the remission or good response should be confirmed based on chest/abdomen/pelvis CT examinations. After obtaining the patient's informed consent to participate in the clinical trial, a brain MRI (MRI-1) will be performed and a baseline assessment of cognitive functions will be carried out using the battery of test listed below.

Patients who at MRI-1 will be diagnosed with cerebral metastasis, depending on the size and number of lesions will be eligible for WBRT (whole brain irradiation) or SRT (brain stereotactic radiotherapy). We propose SRT eligibility treatment criteria as in NSCLC according to the standards of the participating centers. All participating radiotherapy centers must have experience in SRT of brain metastases and up to date radiotherapy equipment suitable for SRT. Subjects who will not have cerebral metastases in the MRI-1 after chemo-radiotherapy will have their next follow-up every 3 months (+/- 2 weeks) up to 2 years, and then every 6 months (+/- 2 weeks) up to 3 years.

At the qualifying visit before MRI-1, and then every 6 months +/- 2 weeks), the patients will have a cognitive examination performed using dedicated neuropsychological tests and QoL assessment using the QLQ-C30 questionnaire. The tests will be conducted in the following order: California verbal learning test (CVLT) with a delay of 15 min, Color connection test (CTT), CVLT (after delay), Benton visual memory test (BNRT), Verbal fluency test by the certified psychologist.

ELIGIBILITY:
Inclusion Criteria:

* confirmed histologically small cell lung cancer, confirmed by staging limited disease SCLC, complete or good response to local chemoradiotherapy, good performance status (ECOG/WHO=0-2), signed informed consent

Exclusion Criteria:

* disseminated disease (ED-SCLC), contraindication to MRI, not able to perform cognitive function tests, poor PS (ECOG/WHO >2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Katedra Onkologii, Wydział Lekarski, Collegium Medicum, Uniwersytet Warmińsko-Mazurski, Olsztyn, Warmia I Mazury, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nawrocki S, Sugajska A. Study protocol: watchful observation of patients with limited small cell lung cancer instead of the PCI-prospective, multi-center one-arm study. BMC Cancer. 2020 Mar 18;20(1):231. doi: 10.1186/s12885-020-06721-8. PMID 32188425